CLINICAL TRIAL: NCT01812343
Title: Mesure de l'Index de Pression Systolique de Cheville après Test d'Effort Maximal.
Brief Title: Value of Ankle Pressure Index After Maximal Exercise Tests
Acronym: VICTOR
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Inclusions objectives raised but patient follow-up reduced to 6 months (impossible to raised secondary objectives)
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PHRC-2011
Record Dates: First submitted 2013-03-04; First posted 2013-03-18 (Estimated); Last update posted 2022-08-02 (Actual); Status verified 2019-11

CONDITIONS: Cardiovascular Diseases
Keywords: Ankle Brachial Index; Maximal Exercise Test
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Exercise Test

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Exercise test (Other): Ankle pressure Index measure before and after Maximal Exercise Tests
  Interventions: Other: Exercise test

INTERVENTIONS:
Other: Exercise test

SUMMARY:
Estimate the response of ankle to brachial pressure index to incremental maximum exercise in subjects free from prior cardiovascular disease.

Estimate morbi-mortality of included patients over a 5 years follow up.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old and more

Exclusion Criteria:

* patient with recent cardiovascular event

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1760 (Actual)
Dates: Start 2009-09-17 (Actual); Primary Completion 2020-05-11 (Actual); Study Completion 2020-05-11 (Actual)

PRIMARY OUTCOMES:
Mean value of post exercise ABI by age categories | up to 15min
  Ankle to brachial index is measured before and after a maximal exercise on a cycle ergometer. results are expressed by age categories of 10 years interval

SECONDARY OUTCOMES:
Prevalence of Morbi-mortality through self completed questionnaires | up to 5 year

CONTACTS AND LOCATIONS:
Overall Officials: Pierre ABRAHAM, PU-PH, Principal Investigator — University Hospital, Angers
Locations (1):
- UHAngers, Angers, France

REFERENCES:
- [Derived] Congnard F, Abraham P, Vincent F, Le Tourneau T, Carre F, Hupin D, Hamel JF, Vielle B, Bruneau A. Ankle to brachial systolic pressure index at rest increases with age in asymptomatic physically active participants. BMJ Open Sport Exerc Med. 2015 Nov 25;1(1):e000081. doi: 10.1136/bmjsem-2015-000081. eCollection 2015. PMID 27900144